CLINICAL TRIAL: NCT06547853
Title: Effect of an Exercise Program on Physical Performance and Health Outcomes in Cancer Survivors
Brief Title: Physical and Health Outcomes With ExeRcise in Cancer SURVIVORS
Acronym: POWERSurviv
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Alagoas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE - 54130721.3.0000.5013
Record Dates: First submitted 2024-07-21; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Female; Exercise
Keywords: Cancer Survivors; Breast Cancer; Physical Exercise
MeSH Terms: conditions — Motor Activity; Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined exercise training (Experimental): In the combined exercise training regimen, participants will perform two hospital-based sessions with 45 minutes of aerobic dance and resistance training. The intensity of the aerobic dance will be ~ 132-135 beats per minute, whereas the intensity of the resistance training will be measured by the subjective rate of perceived exertion. The resistance exercise training regimen was set in a circuit, and participants will perform six exercises per session targeting the large muscle groups. Each exercise will be executed in two sets per session.
  Interventions: Behavioral: Physical exercise

INTERVENTIONS:
Behavioral: Physical exercise — Groups will be enrolled in a 12-week exercise program. The intervention will be carried out in a highly complex oncology center in Maceió-AL, using the FITT components of the prescription: frequency (4 days a week), intensity (aerobic part through musical beats, subjective perception scale and resistance exercises through a number of maximum repetitions), the time of each session will be 45 minutes, the type of activity offered will be combined exercise training and aerobic exercise training (i.e., walking).

SUMMARY:
This study aims to evaluate the effect of a physical exercise intervention model on breast cancer survivors and their adherence. The sample will consist of 30 women with a primary diagnosis of breast cancer. The intervention will be carried out in a highly complex oncology center in Maceió-AL, Brazil, using the FITT components of the prescription: frequency (4 days a week), intensity (aerobic part through musical beats, subjective perception scale and resistance exercises through the number of maximum repetitions), the total time of each session will be 45 minutes. The intervention arms include combined exercise training and aerobic exercise (i.e., walking). Adherence to each intervention evaluated in the 12-week intervention cycle will be measured in each session.

DETAILED DESCRIPTION:
The study participants will be enrolled in a visit to a group of psychologic therapy women cancer survivors who met monthly and who have submitted to breast cancer treatment in a hospital in the city of Maceió (AL), Brazil, classified as High Complexity Oncologic Clinic. At this visit, the proposal for physical exercises will be presented in the hospital area. Volunteers will be scheduled for an in-person visit and assessed for eligibility. Those who meet all the inclusion/exclusion criteria will be invited to integrate the physical exercise intervention.

The 12-week exercise intervention will consist of a combined exercise including an aerobic component (dance) and resistance training, and aerobic exercise (i.e., walking). Participants will be evaluated pre- and post-intervention in terms of several health indicators. All ethical approvals were collected before study initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Women;
2. Adults;
3. confirmed diagnostic of breast cancer and with treatment completed (surgery, radiotherapy, or chemotherapy) within the previous six months.

Exclusion Criteria:

1. present metastatic breast cancer;
2. any clinical condition that would make participating in the exercise intervention impossible.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Exercise adherence | 12-weeks intervention
  Total adherence will be expressed by the percentage of attendance by each participant in the total exercise intervention length. This will be measured by the study staff as the participants presence in each session.

SECONDARY OUTCOMES:
Change in systolic and diastolic blood pressure | 12-weeks
  Blood pressure is going to be measured after 10 minutes in a seated position. Mean Systolic blood pressure and diastolic blood pressure will be evaluated through a digital wrist monitor.
Change in cardiorespiratory fitness | 12-weeks
  cardiorespiratory fitness will be evaluated through the 6-minutes walk test
Change in depression total score | 12-weeks
  Depression will be evaluated using the 9-Item Patient Health Questionnaire (PHQ-9) total score
Change in pain total score | 12-weeks
  Pain will be evaluated using the Brief Pain Inventory (BPI) total score
Change in Health-related Quality of Life total score | 12-weeks
  Health-related quality of life will be evaluated through the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30)
Change in Sleep quality | 12-weeks
  Sleep quality will be evaluated using the The Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Toscano, PhD, Principal Investigator — Federal University of Alagoas Institute of Physical Education and Sports
Locations (1):
- Federal University of Alagoas Institute of Physical Education and Sports, Alagoas, Maceio, Brazil